CLINICAL TRIAL: NCT00810121
Title: Non-inferiority Study of Bi-Profenid® 200 mg Versus Bi-Profenid® 300 mg in Patients Presenting With Pain Related to Closed, Benign, Acute Post-traumatic Conditions of the Motor System or Acute, Non-infectious Rheumatologic Conditions
Brief Title: Study of Non Inferiority Bi-Profenid® 200mg Versus Bi-Profenid® 300mg Among Patients Presenting of the Post-traumatic or Rheumatologic Acute Affections of the Locomotor Apparatus (BIPROPAIN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KETOP_L_03948; 2008-003375-41
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Ketoprofen 100 mg b.i.d. for 5 days
  Interventions: Drug: ketoprofen 100 mg
- 2 (Experimental): Ketoprofen 150 mg b.i.d. for 5 days
  Interventions: Drug: ketoprofen

INTERVENTIONS:
Drug: ketoprofen 100 mg — 100 mg b.i.d. for 5 days
  Arms: 1
Drug: ketoprofen — 150 mg b.i.d. for 5 days
  Arms: 2

SUMMARY:
Primary objective:

To demonstrate the non-inferiority of Bi-Profenid 100 mg x 2 day versus Bi-Profenid 150 mg x 2 day in patients presenting with pain related to closed, benign, acute post-traumatic conditions of the motor system or acute, non-infectious rheumatologic conditions, by comparing, on the one hand, changes in resting pain intensity over the entire day, measured at the end of the day using a numeric scale (NS), over 5 days and, on the other hand, total intake over 5 days of concomitant analgesics.

Secondary Objectives:

* To describe concomitant analgesic treatments
* To describe the time between baseline and use of a step I, II or III analgesic
* To evaluate patients pain relief using a Likert 4-class scale (complete or substantial relief, moderate relief slight relief and absence of relief) at D5
* To evaluate changes in intensity of pain when moving, over the entire day, measured at the end of the day using a numeric scale, over 5 days
* To evaluate the patients overall satisfaction at the end of treatment using a 4-point Simple Verbal Scale (SVS) (very satisfied, somewhat satisfied, somewhat unsatisfied, very unsatisfied)
* To evaluate the patients overall satisfaction at the end of the study using a 4-point Simple Verbal Scale (EVS) (very satisfied, somewhat satisfied, somewhat unsatisfied, very unsatisfied)
* To compare the safety of the two treatments

ELIGIBILITY:
Inclusion criteria :

* Male or female, more than 18 and less than 65 years of age,
* Women using a method of contraception and with a negative pregnancy test before entering the study, or women who have been menopausal for at least 1 year,
* Patients meeting one of the following criteria:
* Closed benign trauma of the motor system occurring within the last 24 hours,
* Contusion of the motor system occurring within the last 24 hours,
* Acute rheumatologic conditions (acute lower back pain, lumbar sciatica, cervicobrachial neuralgia),
* Abarticular rheumatism,
* Requiring treatment with Bi-Profenid for 5 days,
* With resting pain intensity measured on a numeric scale at baseline >or= 3 (before administration of any treatment),
* Receiving a prior medical examination suited to the study

Exclusion criteria :

* Need for surgery,
* Need for hospitalization,
* Need for an analgesic other than step I at the baseline visit,
* Need for treatment with another selective or non-selective NSAID (per os and/or topical), including aspirin, selective cyclo-oxygenase 2 inhibitors, corticosteroids or muscle relaxants at baseline and throughout the study,
* Serious trauma: knee luxation, any fracture, ruptures such as Achilles tendon rupture,
* Sprain treated with a cast,
* Bursitis,
* Local and/or general severe infection,
* Pregnant or nursing women,
* Hypersensitivity to ketoprofen or to any of the excipients of the product,
* Previous history of asthma triggered by taking ketoprofen or substances with similar activity such as other NSAIDs or aspirin,
* Gastrointestinal haemorrhage, cerebrovascular haemorrhage or other active haemorrhage,
* Previous history of digestive haemorrhage or perforation during previous NSAID treatment,
* Active intestinal ulcer,
* Active peptic ulcer, previous history of peptic ulcer or recurrent haemorrhage (2 separate episodes or more of haemorrhage or ulcerations detected),
* Severe hepatic failure,
* Severe renal failure,
* Severe heart failure,
* Uncontrolled hypertension,
* Hypersensitivity or intolerance to gluten, due to the presence of wheat starch (gluten),
* Patients treated with oral anticoagulants, heparins, platelet antiaggregants, selective serotonin reuptake inhibitors (SSRI), lithium, methotrexate, pemetrexed and immunosuppressants

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Resting pain intensity measured using the numeric scale (NS) at the end of the day, and total intake of concomitant analgesics over 5 days. For these two parameters, the maximum value will be assigned to patients who used step II or III analgesics | between D1 and D5, at the end of the day

CONTACTS AND LOCATIONS:
Overall Officials: Marie Sebille, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France